CLINICAL TRIAL: NCT02808325
Title: Prospective Controlled Randomized Double-blind Multicentre Study in Parallel Groups on the Efficacy and Safety of Gelaspan in Combination With Sterofundin ISO in Comparison With Gelofusine in Combination With Sodium Chloride Braun in Patients Scheduled for Abdominal or Pelvic Surgery
Brief Title: Study on the Efficacy and Safety of Gelaspan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: B. Braun Medical LLC (Industry)
Responsible Party: Sponsor
Organization: B. Braun Melsungen AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HC-G-H-1409
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-04

CONDITIONS: Hypovolemia
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- balanced gelatine solution (Experimental): isotonic colloidal volume substitute
  Interventions: Drug: Gelaspan 4%
- non-balanced gelatine solution (Active Comparator): colloidal volume substitute
  Interventions: Drug: Gelofusine 4%

INTERVENTIONS:
Drug: Gelaspan 4% — Gelaspan 4% combined with Sterofundin ISO
  Arms: balanced gelatine solution
Drug: Gelofusine 4% — Gelofusine 4% combined with Sodium Chloride
  Arms: non-balanced gelatine solution

SUMMARY:
It is the objective of the study to investigate the efficacy and safety of two different volume replacement regimens with gelatine solutions.

ELIGIBILITY:
Inclusion:

* Male or female patients ≥ 18 years of age and ≤ 80 years of age.
* Patients scheduled to undergo open elective abdominal or pelvic surgery.
* Anticipated intraoperative volume requirement for gelatine solution is at least 15 mL/kg body weight
* Negative pregnancy test (urine dipsticks) in women of child bearing potential.
* Provision of voluntary consent to participate in the study, following a full explanation of the nature and purpose of the study, by signing the informed consent form approved by the regulatory authorities of the Russian Federation and Local Ethics Committee (LEC) prior to all evaluations.

Exclusion:

* Patients of ASA-class > III.
* Known hypersensitivity to gelatine or to any of the constituents of the solution.
* Patients treated with other colloid solutions and / or blood products 24 hours prior to surgery.
* Patients on hemodialysis.
* Patients suffering from:

  * Decompensated renal function (i.e. serum creatinine > 3.0 mg/dL)
  * Hypervolemia;
  * Severe heart failure;
  * Moderate lung edema;
  * Hyperhydration;
  * Severe blood coagulation disorders (aPTT >2.5 x ULN or fibrinogen < 0.5 x LLN or INR >2.5 x ULN);
  * Hypernatremia (serum Na+ > 150 mmol/L);
  * Hyperchloremia (serum Cl- > 110 mmol/L);
  * Hypercalcemia (serum ionized Ca++ > 1.5 mmol/L);
  * Metabolic alkalosis;
  * Severe generalized edema;
  * Intracranial haemorrhage;
  * Hyperkalemia (serum K+ > 5.5 mmol/L).
* Pregnancy and/or nursing.
* Hypertension with the Systolic Blood Pressure > 180 mm Hg and Diastolic Blood Pressure > 110 mm Hg identified at screening.
* Patients who in the investigator's opinion couldn't take part in the study.
* Simultaneous participation in another clinical trial.
* Emergencies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-06; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Base Excess | Change in base excess from baseline to end of surgery

SECONDARY OUTCOMES:
Base Excess | Change in base excess from baseline to 12 hours after end of surgery
Adverse events | until 12 hours after end of surgery
Hemodynamics | until 12 hours after end of surgery
Renal Function | until 12 hours after end of surgery
Arterial blood gas analysis | until 12 hours after end of surgery
Coagulation status | until 12 hours after end of surgery

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - Road Clinical Hospital of JSC "Russian Railways, Saint Petersburg
  - North-Western Federal Medical Research Center n.a. V.A. Almazov, Saint Petersburg
  - City Clinical Oncology Dispensary, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No